CLINICAL TRIAL: NCT05078879
Title: A Phase 1 Study of Empagliflozin as Treatment for Severe Congenital Neutropenia Due to G6PC3 Deficiency
Brief Title: Empagliflozin as a Treatment for Severe Congenital Neutropenia Due to G6PC3 Deficiency
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 10000236; 000236-I
Record Dates: First submitted 2021-10-14; First posted 2021-10-15 (Actual); Last update posted 2025-06-26 (Actual); Status verified 2025-06

CONDITIONS: Crohn's Disease; Glycogen Metabolism; Inflammatory Bowel Disease (IBD)
Keywords: Glycogen metabolism; Jardiance; Inflammatory Bowe Disease (IBD); G6PT deficiency; 1,5-AG
MeSH Terms: conditions — Crohn Disease; Inflammatory Bowel Diseases | interventions — empagliflozin

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment Arm (Experimental): Patients with GCPC3 will receive daily Empagliflozin for 12 months.
  Interventions: Drug: Empagliflozin

INTERVENTIONS:
Drug: Empagliflozin — This is an open-label pilot study to evaluate the efficacy, safety, and tolerability of empagliflozin as a treatment for severe congenital neutropenia (SCN) in patients with glucose-6-phosphatase 3 (G6PC3) deficiency. Participants will be on a 12-month daily regimen of empagliflozin at a starting dose of 10 mg (phase A), which may be increased after 2 months to 25 mg (phase B). Evaluate the safety and efficacy of the biomarker response (the change in absolute neutrophil count [ANC] after one year of empagliflozin treatment relative to baseline ANC prior to drug treatment) in patients with G6PC3 deficiency.

SUMMARY:
Background:

Severe congenital neutropenia (SCN) is an immune system disease. People with SCN do not have enough of a kind of white blood cell called neutrophils. This means they get sick easily from infections. Some drugs to treat SCN have lots of side effects. Researchers want to see if a the drug empagliflozin can help increase the number of neutrophils in a person with SCN.

Objective:

To see if a drug called empagliflozin can help people with SCN.

Eligibility:

Adults aged 18 and older with SCN.

Design:

Participants will be screened with a physical exam, medical history, and blood tests. They may have a pregnancy test.

Participants will have study visits and local lab visits. They will repeat the screening tests. They will have heart and lung function tests. They will have an ultrasound of the liver and spleen. Their skin symptoms will be photographed. They may have consultations with specialists. They may give a stool sample. They may have an optional colonoscopy with tissue sample collection. They may have an optional bone marrow biopsy and aspirate. They may have an optional magnetic resonance imaging scan of their heart.

Participants will be admitted to NIH for 5 7 days. They will start taking the study drug as a pill once daily. They will be monitored for side effects.

Participants will take the study drug at home for 12 months. They will use a fingerstick blood glucose meter to measure blood sugar at home.

Participants may be able to take the study drug through their local doctor after the study ends.

Participation will last for 15 months.

DETAILED DESCRIPTION:
One symptom of G6PC3 deficiency is recurrent infections resulting from severe congenital neutropenia (SCN). Data suggest that SCN is the result of accumulation of the toxic dietary metabolite 1,5 anhydroglucitol 6 phosphate (1,5-AG6P) in leukocytes. This buildup inhibits glycolytic metabolism, thus impairing their function. Increasing urinary glucose excretion results in the urinary excretion of the precursor to 1,5-AG6P, and will likely reduce levels of 1,5-AG6P in leukocytes.

In this phase 1 open-label study, we will evaluate the safety, tolerability, and efficacy of the sodium glucose co transporter 2 inhibitor empagliflozin in patients with G6PC3 deficiency. Empagliflozin is FDA approved in doses of 10 or 25 mg daily for treatment of type 2 diabetes in adults. Eligible participants (n=5) aged >=18 years will be on a 2-month daily regimen of 10 mg of oral empagliflozin (phase A). Participants may then be increased to 25 mg daily (phase B) if the participant fails to achieve an adequate improvement in neutropenia during phase A and is able to tolerate the higher dose, or alternatively may continue on the 10-mg dose. Participants will temporarily discontinue any current granulocyte colony-stimulating factor (G-CSF) regimen starting at least 7 days before the empagliflozin regimen begins, to remove or reduce the effects of concomitant G-CSF so the baseline ANC can be evaluated without confounding factors.

During phase A, participants will have blood drawn locally every two weeks for clinical lab evaluations (including ANC). A member of the study team will also contact the participant for remote AE assessment at each blood draw. During phase B, blood draws and remote AE assessments will be monthly for the first 4 months, and bimonthly for the last 6 months. Participants will have outpatient study visits at the NIH Clinical Center at the end of phase A (month 2), and at months 6 and 12 during phase B.

ELIGIBILITY:
* INCLUSION CRITERIA:

  1. Aged >=18 years.
  2. Documented SCN due to G6PC3 deficiency defined by genetic testing.
  3. History of ANC consistently <1000 cells/microL when not treated with G-CSF.
  4. Current ANC<1000 cells/microL when not treated with G-CSF.
  5. Participants must agree not to become pregnant for the duration of the study. Study participants must use 2 methods of birth control when engaging in sexual activities that can result in pregnancy, beginning 30 days before the first dose of empagliflozin through one month after treatment ends. One method must be a male or female condom. The other method may be any of the following:

     1. Hormonal contraception.
     2. Diaphragm or cervical cap with a spermicide.
     3. Intrauterine device.
  6. Able to provide informed consent.

EXCLUSION CRITERIA:

Individuals meeting any of the following criteria will be excluded from study participation:

1. Renal failure or eGFR<45 mL/min/1.73 m^2.
2. Type 1 diabetes mellitus.
3. Fasting hypoglycemia (<60 mg/dL).
4. Known hypersensitivity or allergy to any component of empagliflozin.
5. Pregnant.
6. Breastfeeding.
7. Any condition that, in the opinion of the investigator, contraindicates participation in this study.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2021-11-16 (Actual); Primary Completion 2025-05-02 (Actual); Study Completion 2025-05-21 (Actual)

PRIMARY OUTCOMES:
Absolute Neutrophil Count | End of Treatment at 12 months
  ANC increase by >500 cells/uL over baseline (measured at least 3x over 2 days)
Safety | End of Treatment at 12 months
  No Grade 3/4 toxicities that require pause of the study drug.

SECONDARY OUTCOMES:
Neutrophil Function | End of Treatment at 12 months
  Improved in vitro NADPH oxidase function, Staphylococcus aureus killing assay, and chemotaxis assay.

CONTACTS AND LOCATIONS:
Overall Officials: David H McDermott, M.D., Principal Investigator — National Institute of Allergy and Infectious Diseases (NIAID)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Banka S, Newman WG. A clinical and molecular review of ubiquitous glucose-6-phosphatase deficiency caused by G6PC3 mutations. Orphanet J Rare Dis. 2013 Jun 13;8:84. doi: 10.1186/1750-1172-8-84. PMID 23758768
- [Background] Dale DC, Bolyard AA, Marrero T, Kelley ML, Makaryan V, Tran E, Leung J, Boxer LA, Kishnani PS, Austin S, Wanner C, Ferrecchia IA, Khalaf D, Maze D, Kurtzberg J, Zeidler C, Welte K, Weinstein DA. Neutropenia in glycogen storage disease Ib: outcomes for patients treated with granulocyte colony-stimulating factor. Curr Opin Hematol. 2019 Jan;26(1):16-21. doi: 10.1097/MOH.0000000000000474. PMID 30451720
- [Background] Boztug K, Appaswamy G, Ashikov A, Schaffer AA, Salzer U, Diestelhorst J, Germeshausen M, Brandes G, Lee-Gossler J, Noyan F, Gatzke AK, Minkov M, Greil J, Kratz C, Petropoulou T, Pellier I, Bellanne-Chantelot C, Rezaei N, Monkemoller K, Irani-Hakimeh N, Bakker H, Gerardy-Schahn R, Zeidler C, Grimbacher B, Welte K, Klein C. A syndrome with congenital neutropenia and mutations in G6PC3. N Engl J Med. 2009 Jan 1;360(1):32-43. doi: 10.1056/NEJMoa0805051. PMID 19118303
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_000236-I.html